CLINICAL TRIAL: NCT05876728
Title: Role of Irisin/FNDC5 (rs3480) Single Nucleotide Polymorphism in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Badway Hemdan, lecturer of medical biochemistry, Sohag University
Other Study IDs: Soh-Med-23-04-10PD
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group: 50 patient of histologically confirmed breast cancer
  Interventions: Genetic: Genotyping
- control group: 50 healthy volunteers with no clinical evidence of any neoplastic disorder
  Interventions: Genetic: Genotyping

INTERVENTIONS:
Genetic: Genotyping — Genotyping of rs 3480 of irisin gene using the Taqman Allelic Discrimination assay technique.

SUMMARY:
Breast cancer is the most frequent cancer in women worldwide. Its incidence is increasing but mortality has decreased in a considerable way due to the combined effect of early detection and improvement in treatment .

Irisin is encoded by the FNDC5 gene, whose expression is controlled by the peroxi- some proliferator activated receptor gamma coactivator 1 alpha (PGC-1α). PGC-1α is a transcriptional co-activator which does not bind directly to DNA. Studies indicated that the estrogen-related receptor alpha (ERRα) could be a factor that plays a role in PGC-1α binding to DNA. ERRα is encoded by the ESRRA gene and is an orphan nuclear receptor, which has two domains. One of them allows the interaction with DNA, and the second one with a ligand. The ERRα structure is similar to that of the estrogen receptor alpha (ERα), but this receptor does not bind to natural estrogens. ERRα interacts with a canonical sequence of the estrogen response elements (ERRE). ERRα and ERα could compete with each other to bind to similar DNA elements. Together, ERRα binds to DNA, in complex with PGC-1α, to regulate the activity of genes such as FNDC5 .

CA15-3, a high molecular weight glycoprotein (300-450 kDa), is produced by the epithelial ducts and acinic breast cells and is then secreted in milk normally. It has been widely used for the prediction of bone metastases in patients with breast cancer .

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed breast cancer

Exclusion Criteria:

* • History of other tumors.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A Case control study will be conducted on 100 patients with histologically confirmed breast cancer, and a control group of 50 healthy volunteers with no clinical evidence of any neoplastic disorder.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
find a possible association between irisin gene single nucleotide polymorphism with breast cancer | 12 months
  - find a possible association between irisin gene single nucleotide polymorphism with breast cancer risk and the distribution of its alleles, in relation to many clinical parameters of the cancer group.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peto R, Boreham J, Clarke M, Davies C, Beral V. UK and USA breast cancer deaths down 25% in year 2000 at ages 20-69 years. Lancet. 2000 May 20;355(9217):1822. doi: 10.1016/S0140-6736(00)02277-7. No abstract available. PMID 10832853
- [Background] Balmain A, Gray J, Ponder B. The genetics and genomics of cancer. Nat Genet. 2003 Mar;33 Suppl:238-44. doi: 10.1038/ng1107. PMID 12610533
- [Background] Nowinska K, Jablonska K, Ciesielska U, Piotrowska A, Haczkiewicz-Lesniak K, Pawelczyk K, Podhorska-Okolow M, Dziegiel P. Association of Irisin/FNDC5 with ERRalpha and PGC-1alpha Expression in NSCLC. Int J Mol Sci. 2022 Nov 17;23(22):14204. doi: 10.3390/ijms232214204. PMID 36430689
- [Background] Fakhari A, Gharepapagh E, Dabiri S, Gilani N. Correlation of cancer antigen 15-3 (CA15-3) serum level and bony metastases in breast cancer patients. Med J Islam Repub Iran. 2019 Dec 19;33:142. doi: 10.34171/mjiri.33.142. eCollection 2019. PMID 32280648